CLINICAL TRIAL: NCT00059943
Title: Pharmacokinetics of Weekly Docetaxel in Patients Age 65 and Older With Metastatic Breast or Lung Cancer
Brief Title: Docetaxel in Treating Older Patients With Metastatic Breast, Lung, or Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 01-136; MSKCC-01136
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer; Lung Cancer; Prostate Cancer
Keywords: stage IV breast cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; recurrent breast cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

INTERVENTIONS:
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well docetaxel works in treating older patients with metastatic breast, lung, or prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the pharmacokinetics of docetaxel in older patients with metastatic breast, lung, or prostate cancer.
* Determine the response of patients treated with this drug.
* Determine the toxicity of this drug in these patients.
* Determine the short-term changes in functional status, in terms of activities of daily living, independent activities of daily living, and Karnofsky performance status, in patients treated with this drug.
* Correlate the number of comorbid conditions at baseline with declines in functional status in patients treated with this drug.

OUTLINE: Patients receive docetaxel IV over 30 minutes once weekly for 3 weeks. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven metastatic breast, lung, or prostate cancer
* Measurable disease
* No untreated CNS metastases
* No symptomatic CNS metastases requiring escalating doses of corticosteroids
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 65 and over

Sex

* Not specified

Menopausal status

* Not specified

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Hemoglobin at least 8.0 g/dL
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin normal
* SGOT and/or SGPT no greater than 2.5 times upper limit of normal (ULN) with alkaline phosphatase no greater than ULN OR
* Alkaline phosphatase no greater than 4 times ULN with SGOT and SGPT no greater than ULN

Renal

* Not specified

Cardiovascular

* No history of cardiac arrhythmia
* No congestive heart failure
* No myocardial infarction within the past 6 months

Other

* No prior severe hypersensitivity reaction to docetaxel or other drugs containing polysorbate 80
* No allergy to macrolide antibiotics
* No grade 2 or greater peripheral neuropathy
* No concurrent serious or uncontrolled infection
* Able to read, write, and converse in English

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Recovered from prior chemotherapy

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* Recovered from prior radiotherapy

Surgery

* Not specified

Other

* No concurrent CYP3A4-inducing or inhibiting medications or herbal remedies
* No concurrent grapefruit juice
* No concurrent ethanol

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 2002-09; Primary Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of docetaxel

SECONDARY OUTCOMES:
Correlation between docetaxel clearance with estimated cytochrome p450 activity by the Erythromycin Breath Test
Response
Toxicity
Correlation between toxicity and functional status decline
Relationship between comorbid conditions at baseline and declines in functional status

CONTACTS AND LOCATIONS:
Overall Officials: Arti Hurria, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States